CLINICAL TRIAL: NCT03294382
Title: Botulinum Toxin to Improve Results in Epicanthoplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ru-Lin Huang, Ph.D., M.D., Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9hospital
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Scar; Intercanthal Distance Ratio
Keywords: epicanthoplasty; Botulinum Toxins; scar; intercanthal distance; blepharoplasty
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin (Experimental): 5U Botulinum toxin in 0.1 mL normal saline, administered in one of the intercanthus
  Interventions: Drug: Botulinum toxin type A
- Normal Saline (Placebo Comparator): 0.1 mL normal saline, administered in the other intercanthus
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin type A — 5U botulinum toxin in 0.1 mL normal saline, injected in two points at one side, 2.5U per point, local injection
  Arms: Botulinum toxin
Drug: Placebo — 0.1 mL normal saline, injected in two points at one side, 0.05 mL per point, local injection
  Arms: Normal Saline

SUMMARY:
Medial epicanthal fold is a common skin fold in the inner part of the eye in more than 50% Asia population, giving the illusion of a shorter palpebral fissure length and a wider intercanthal distance. Currently, various epicanthoplasty techniques have been well described to correct epicanthus fold. However, hypertrophic scarring after epicanthoplasty remains a clinical challenge, which seems inevitable and may leading to unpleasing supratarsal crease, recurrence of medial epicanthus fold, even obvious scar formation. Botulinum toxin type A (BTX-A) is widely used for facial rejuvenation and many other medical indications. It is a potent neurotoxin that indirectly blocks neuromuscular transmission and leads to functional denervation of striated muscle for 2 to 6 months after injection. Recently, experimental study and clinical trails have revealed that BTX-A can inhibit the growth of fibroblasts derived from hypertrophic scars and influenced the expression of transforming growth factor-β1. Therefore, we hypothesized that BTX-A can improve hypertrophic scarring after epicanthoplasty through release orbicularis oculi muscle tension, inhibit fibroblast growth, and reduce collagen production. The main aim of this trail is to evaluate the efficiency of BTX-A injection on improving hypertrophic scaring after epicanthoplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe congenital epicanthus.
* patients accept Park Z epicanthoplasty.
* Written informed consent given

Exclusion Criteria:

* epicanthus caused by trauma, surgical injury.
* patients with both epicanthus and blepharopotosis.
* patients with blepharophimosis-ptosis-epicanthus inversus syndrome, or only inversus epicanthus
* patients underwent Botulinum Toxin Type A periocular injection within 6 months
* patients ever have been allergic to Botulinum Toxin Type A or any components of Botulinum Toxin Type A

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar scale | 6 month
  Vancouver scar scale measures pigmentation, vascularity, pliability and scar height on the postoperative 6 month F/U
intercanthal distance ratio | 6 month
  the ratio of the intercanthal distance to the interpupillary distance

SECONDARY OUTCOMES:
Photographic measurement | 6 month
  The scar width of the patient's picture at 6 month after surgery will be measured using photoshop CS3 extended. One ruler will be placed on the patient's nose before taken the photo. Then the scar width could be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Ru-Lin Huang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair: a double-blinded, randomized, vehicle-controlled clinical trial. PLoS One. 2014 Dec 26;9(12):e115690. doi: 10.1371/journal.pone.0115690. eCollection 2014. PMID 25541942
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair. Plast Reconstr Surg. 2014 Sep;134(3):511-516. doi: 10.1097/PRS.0000000000000416. PMID 25158709
- [Background] Al-Qattan MM, Al-Shanawani BN, Alshomer F. Botulinum toxin type A: implications in wound healing, facial cutaneous scarring, and cleft lip repair. Ann Saudi Med. 2013 Sep-Oct;33(5):482-8. doi: 10.5144/0256-4947.2013.482. PMID 24188943
- [Background] Zelken J, Yang SY, Chang CS, Chang CJ, Yang JY, Chuang SS, Chen HC, Hsiao YC. Donor Site Aesthetic Enhancement With Preoperative Botulinum Toxin in Forehead Flap Nasal Reconstruction. Ann Plast Surg. 2016 Nov;77(5):535-538. doi: 10.1097/SAP.0000000000000625. PMID 26418784
- [Background] Kim YS, Lee HJ, Cho SH, Lee JD, Kim HS. Early postoperative treatment of thyroidectomy scars using botulinum toxin: a split-scar, double-blind randomized controlled trial. Wound Repair Regen. 2014 Sep-Oct;22(5):605-12. doi: 10.1111/wrr.12204. Epub 2014 Aug 26. PMID 24898579
- [Result] Kwon B, Nguyen AH. Reconsideration of the Epicanthus: Evolution of the Eyelid and the Devolutional Concept of Asian Blepharoplasty. Semin Plast Surg. 2015 Aug;29(3):171-83. doi: 10.1055/s-0035-1556849. PMID 26306084
- [Result] Elhefnawy AM. Assessment of intralesional injection of botulinum toxin type A injection for hypertrophic scars. Indian J Dermatol Venereol Leprol. 2016 May-Jun;82(3):279-83. doi: 10.4103/0378-6323.173586. PMID 27088929
- [Result] Shaarawy E, Hegazy RA, Abdel Hay RM. Intralesional botulinum toxin type A equally effective and better tolerated than intralesional steroid in the treatment of keloids: a randomized controlled trial. J Cosmet Dermatol. 2015 Jun;14(2):161-6. doi: 10.1111/jocd.12134. Epub 2015 Mar 24. PMID 25810045
- [Result] Robinson AJ, Khadim MF, Khan K. Keloid scars and treatment with Botulinum Toxin Type A: the Belfast experience. J Plast Reconstr Aesthet Surg. 2013 Mar;66(3):439-40. doi: 10.1016/j.bjps.2012.08.042. Epub 2012 Oct 23. No abstract available. PMID 23092904
- [Result] Zhang DZ, Liu XY, Xiao WL, Xu YX. Botulinum Toxin Type A and the Prevention of Hypertrophic Scars on the Maxillofacial Area and Neck: A Meta-Analysis of Randomized Controlled Trials. PLoS One. 2016 Mar 17;11(3):e0151627. doi: 10.1371/journal.pone.0151627. eCollection 2016. PMID 26985661
- [Derived] Huang RL, Ho CK, Tremp M, Xie Y, Li Q, Zan T. Early Postoperative Application of Botulinum Toxin Type A Prevents Hypertrophic Scarring after Epicanthoplasty: A Split-Face, Double-Blind, Randomized Trial. Plast Reconstr Surg. 2019 Oct;144(4):835-844. doi: 10.1097/PRS.0000000000006069. PMID 31568286